CLINICAL TRIAL: NCT04376658
Title: Assessment of Health-related Quality of Life and Long-term Outcomes After Hospitalization for COVID-19: A Multicenter Prospective Cohort Study
Brief Title: Quality of Life and Long-term Outcomes After Hospitalization for COVID-19
Status: Completed | Type: Observational
Sponsor: Hospital Moinhos de Vento (Other)
Collaborators: Hospital Israelita Albert Einstein (Other); Hospital Sirio-Libanes (Other); Hospital do Coracao (Other); Hospital Alemão Oswaldo Cruz (Other); Beneficência Portuguesa de São Paulo (Other); Brazilian Clinical Research Institute (Other); Brazilian Research In Intensive Care Network (Network)
Responsible Party: Sponsor
Other Study IDs: Coalition COVID-19: Long-term
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Quality of Life; Long-term Outcomes; Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cohort 1 (Coalition I): Adult hospitalized patients with proven or suspected SARS-Cov-2 infection with up to 4L/minute oxygen supply through nasal catheter.
  Interventions: Other: COVID-19 Severity
- Cohort 2 (Coalition II): Adult hospitalized patients with proven or suspected SARS-Cov-2 infection needing oxygen supplementation > 4L/min on nasal catheter or HFNC or NIV or MV or ECMO.
  Interventions: Other: COVID-19 Severity
- Cohort 3 (Coalition III): Adult hospitalized patients with proven or suspected SARS-Cov-2 infection with moderate or severe ARDS according to the Berlin definition
  Interventions: Other: COVID-19 Severity
- Cohort 4 (Coalition IV): Adult hospitalized patients with proven SARS-Cov-2 infection and D-dimer above the upper limit of the normal range
  Interventions: Other: COVID-19 Severity
- Cohort 5 (Coalition VI): Adult hospitalized patients with proven SARS-Cov-2, needing oxygen supplementation to maintain SpO2 > 93%, and two or more of the following inflammatory tests: D-dimer > 1,000 ng/mL; C reactive protein (CRP) > 5 mg/dL; Ferritin > 300 mg/dL; Lactate dehydrogenase (LDH) > upper limit of normal
  Interventions: Other: COVID-19 Severity

INTERVENTIONS:
Other: COVID-19 Severity — Disease severity characterized by the highest six-level ordinal scale during the hospital stay, which consists of the following categories: a score of 1 indicated not hospitalized; 2, hospitalized and not receiving supplemental oxygen; 3, hospitalized and receiving supplemental oxygen; 4, hospitalized and receiving oxygen supplementation administered by a high-flow nasal cannula or noninvasive ventilation; 5, hospitalized and receiving mechanical ventilation; and 6, death

SUMMARY:
The present study aims to assess the determinants of health-related quality of life and long-term outcomes among survivors of hospitalization for Covid-19 in Brazil. The investigators will conduct a multicenter prospective cohort study nested in randomized clinical trials (coalition Covid-19 Brazil initiative) originally designed to assess the effects of specific Covid-19 treatments. Adult survivors of hospitalization due to proven or suspected SARS-CoV-2 infection will be followed up for a period of one year by means of structured telephone interviews. The primary outcome is one-year health-related quality of life assessed by the EQ-5D-3L. Secondary outcomes include all-cause mortality, rehospitalizations, return to work or study, physical functional status assessed by the Lawton & Brody Instrumental Activities of Daily Living Scale, dyspnea assessed by the modified medical research council dyspnea scale, need of long-term ventilatory support, symptoms of anxiety and depression assessed by the Hospital Anxiety and Depression Scale, and symptoms of posttraumatic stress disorder assessed by the Impact of Event Scale-revised.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Hospitalization due to proven or suspected SARS-CoV-2 infection
* Meeting eligibility criteria for Coalition Covid-19 Brazil randomized clinical trials

Exclusion Criteria:

* Death during the hospitalization
* Absence of telephone contact
* Absence of proxy for patients with communication difficulties
* Refusal or withdrawal of agreement to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult survivors of hospitalization due to proven or suspected SARS-CoV-2 infection
Sampling Method: Non-Probability Sample
Enrollment: 1508 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
One-year utility score of health-related quality of life | The outcome will be assessed 12 months after enrollment.
  The outcome will be assessed using the Brazilian version of the Euroqol-5D-3L (EQ-5D3L) questionnaire. The utility score derived from the EQ5D-3L ranges from 0 (death) to 1 (perfect health).

SECONDARY OUTCOMES:
Incidence of all-cause mortality | The outcome will be assessed 3, 6, 9 and 12 months after enrollment.
  Incidence of all-cause mortality.
Incidence of rehospitalizations | The outcome will be assessed 3, 6, 9 and 12 months after enrollment.
  Incidence of all-cause rehospitalizations.
Percentage of return to work or study | The outcome will be assessed 3, 6, 9 and 12 months after enrollment.
  Percentage of return to work or study among patients that were working or studying at the moment of hospitalization.
Score of Instrumental Activities of Daily Living | The outcome will be assessed 3, 6, 9 and 12 months after enrollment.
  The outcome will be assessed using the Lawton & Brody Instrumental Activities of Daily Living Scale (the score ranges from 0 to 8, with higher scores indicating less dependence).
Score of dyspnea | The outcome will be assessed 3, 6, 9, and 12 months after enrollment.
  The outcome will be assessed using the modified medical research council dyspnea scale. Scores ranges from 0 to 4, with higher scores indicating worse symptoms.
Percentage of long-term ventilatory support need | The outcome will be assessed 3, 6, 9 and 12 months after enrollment.
  Percentage of patients requiring oxygen therapy, non-invasive ventilation, or mechanical ventilation.
Symptoms of anxiety and depression | The outcome will be assessed 3, 6, 9 and 12 months after enrollment.
  The outcome will be assessed using the Hospital Anxiety and Depression Scale (anxiety and depression scores range from 0 to 21, with higher scores indicating worse symptoms).
Symptoms of posttraumatic stress disorder | The outcome will be assessed 3, 6, 9 and 12 months after enrollment.
  The outcome will be assessed using the Impact Event Scale-Revised (the score ranges from 0 to 88, with higher scores indicating worse symptoms).
Utility score of health-related quality of life at 3, 6, and 9 months | The outcome will be assessed 3, 6, and 9 months after enrollment.
  The outcome will be assessed using the Brazilian version of the Euroqol-5D-3L (EQ-5D3L) questionnaire. The utility score derived from the EQ5D-3L ranges from 0 (death) to 1 (perfect health).
Score of self-rated health | The outcome will be assessed 3, 6, 9, and 12 months after enrollment.
  The outcome will be assessed using the visual analogue scale of the Brazilian version of the Euroqol-5D-3L questionnaire (EQ-VAS; score range from o to 100, with higher scores indicating better self-rated health).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
The authors encourage interested parties to contact the corresponding author with data sharing requests, including for access to additional unpublished data.

REFERENCES:
- [Background] Rosa RG, Robinson CC, Veiga VC, Cavalcanti AB, Azevedo LCP, Machado FR, Berwanger O, Avezum A, Lopes RD, Lisboa TC, Teixeira C, Zampieri FG, Tomazini BM, Kawano-Dourado L, Schneider D, Souza D, Santos RDRMD, Silva SSD, Trott G, Gimenes BDP, Souza AP, Barroso BM, Costa LS, Brognoli LG, Pelliccioli MP, Studier NDS, Schardosim RFC, Haubert TA, Pallaoro VEL, Oliveira DM, Velho PI, Medeiros GS, Gazzana MB, Zavascki AP, Pitrez PM, Oliveira RP, Polanczyk CA, Nasi LA, Hammes LS, Falavigna M. Quality of life and long-term outcomes after hospitalization for COVID-19: Protocol for a prospective cohort study (Coalition VII). Rev Bras Ter Intensiva. 2021 Jan-Mar;33(1):31-37. doi: 10.5935/0103-507X.20210003. PMID 33886851
- [Derived] Rosa RG, Cavalcanti AB, Azevedo LCP, Veiga VC, de Souza D, Dos Santos RDRM, Schardosim RFC, Rech GS, Trott G, Schneider D, Robinson CC, Haubert TA, Pallaoro VEL, Brognoli LG, de Souza AP, Costa LS, Barroso BM, Pelliccioli MP, Gonzaga J, Studier NDS, Dagnino APA, Neto JM, da Silva SS, Gimenes BDP, Dos Santos VB, Estivalete GPM, Pellegrino CM, Polanczyk CA, Kawano-Dourado L, Tomazini BM, Lisboa TC, Teixeira C, Zampieri FG, Zavascki AP, Gersh BJ, Avezum A, Machado FR, Berwanger O, Lopes RD, Falavigna M. Association between acute disease severity and one-year quality of life among post-hospitalisation COVID-19 patients: Coalition VII prospective cohort study. Intensive Care Med. 2023 Feb;49(2):166-177. doi: 10.1007/s00134-022-06953-1. Epub 2023 Jan 3. PMID 36594987
- See also: Study Protocol — https://pubmed.ncbi.nlm.nih.gov/33886851/